CLINICAL TRIAL: NCT07124403
Title: Evaluation of the Pre-therapeutic Activity of Dihydropyrimidine dEShydrogenase (DPD) in Patients With Cancer and/or Renal Failure
Brief Title: DESIR. Evaluation of the Pre-therapeutic Activity of Dihydropyrimidine dEShydrogenase (DPD) in Patients With Cancer and/or Renal Failure
Acronym: DESIR
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/907
Record Dates: First submitted 2025-07-04; First posted 2025-08-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Renal Impairment; Digestive Cancers; Breast Cancer
MeSH Terms: conditions — Renal Insufficiency; Gastrointestinal Neoplasms; Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENT WITH SOLID TUMOR OR RENAL IMPAIRMENT
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — DPD Activity wil be assessed from blood samples
Diagnostic Test: Blood sampling — Measurement of uracilemia and assessment of renal function

SUMMARY:
Fluoropyrimidine drugs (5-Fluorouracil or 5-FU and its prodrug capecitabine) are a widely used in the treatment of numerous solid tumors in adults. Approximately 85% of administered 5-FU is rapidly catabolized in the liver into inactive dihydrofluorouracil (5-FUH2) by dihydro-pyrimidine dehydrogenase (DPD), leaving only a small fraction of the initial drug for an eventual transformation into cytotoxic metabolites. Impeded DPD activity is associated to an increase of cytotoxic metabolites leading to potentially very severe toxicities.

To prevent these toxicities, a pre-therapeutic measurement of plasma uracil can help assess DPD activity. Indeed, uracil is an endogenous substrate of DPD and an increase in its plasma concentration may be associated with a decrease in DPD activity. In this case, a reduction of the fluoropyrimidine dose is suggested.

However, the investigators observed that uracilemia increased concomitantly to the severity of renal impairment. There are two possible explanations for this observation. Either the renal impairment reduces the renal elimination of uracil from blood, or DPD activity is actually impaired. In both cases, this can explain an increase in plasma uracil concentration.

However, the impact on fluoropyrimidine dosage is different in the two cases. If the increase in uracilemia is due to renal impairment, DPD activity remains unaffected and there is no need to reduce the fluoropyrimidine dose. If DPD activity is actually impaired, a reduction in the fluoropyrimidine dose is required. In cases of renal impairment, uracilemia may therefore not be as relevant for DPD assessment as in the absence of renal impairment.

To assess if DPD activity is actually impede during renal impairment, the DPD activity of Peripheral Blood Mononuclear Cells (PBMCs) will be assessed together with uracilemia in patients with or without renal impairment. As uracilemia decreases after dialysis, the DPD activity of Peripheral Blood Mononuclear Cells (PBMCs) will also be assessed in patient before and after dialysis. Four groups of 50 patients will be studied: patients with normal renal function with hyperuracilemia (uracilemia ≥ 16 ng/mL) or normal uracilemia (uracilemia < 16 ng/mL) ; and patients with renal impairment with hyperuracilemia (uracilemia ≥ 16 ng/mL) or normal uracilemia (uracilemia < 16 ng/mL).

The main objective of the study is to describe the distribution of DPD activity in these four populations. The secondary objectives are to determine in normorenal patients the optimal threshold for DPD activity in non-deficient patients, allowing differentiation between deficient and non-deficient patients based on uracilemia ; and to describe in patients with impaired renal function the distribution of uracilemia with respect to the threshold previously described with the aim of verifying the relevance of uracilemia as a marker of DPD activity in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Affiliation to the Social Security System
* Patients with breast or digestive cancer for whom a fluoroptmidine therapy is being considered
* OR Patients on dialysis (GFR < 10 ml/min/1.73 m²)
* OR Nephrology patients with IR

Exclusion Criteria:

* Patient with anemia < 8.5 g/dl
* Patient with LDH > 2 x > ULN
* Legal incapacity or limited legal capacity
* Subject without health insurance
* Subject in the exclusion period of another study or in the "national volunteer file"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with breast or digestive cancer patients on dialysis patients with IR
Sampling Method: Probability Sample
Enrollment: 742 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
DPD Activity measurement in blood | 3 years
  DPD Activity is assessed in PBMC in µmole of 5FUH2 / h / 1 million cells
Uracilemia in plasma | 3 years
  Uracilemia will be measured in plasma in µg/L
uracilemia-based DPD activity measurement | 3 years
  differentiation between deficient and non-deficient patients will be based on uracilemia (<16, ≥16)
assessment of renal function using eGFR | 3 years
  eGFR is expressed in ml/min/1.73m²
sex | 3 years
  M/F used for eGFR calculation
Age | 3 years
  Years, used for eGFR calculation
creatininemia | 3 years
  µmol/l, used for eGFR calculation